CLINICAL TRIAL: NCT05643261
Title: Can a Strength and Technique Intervention Reduce Knee Abduction Moment in Young Female Handball Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Norges idrettshøgskole (Other)
Responsible Party: Principal Investigator, Tron Krosshaug, Professor Tron Krosshaug PhD, Norges idrettshøgskole
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Søknad 233 - 160622
Record Dates: First submitted 2022-11-21; First posted 2022-12-08 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: ACL Injury
Keywords: ACL injury prevention; Biomechanics; Sidestep cutting; Strength training
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: All players in the intervention group will complete the targeted muscle and technique training integrated into their handball training, while players in the control group only continue their regular handball training. There will be a training of the coaches on site, who assess the training of the intervention group during the entire period and document the participation of the players accordingly.The strength training consists of three exercises (clam shell, side plank, calf raises) with an progressive overload after two to three weeks to ensure a continuous muscle stimulation. The technique training consists of different cutting variations with a focus on forefoot landings and conscious control of the knee to avoid high knee valgus movement and KAM respectively.
Masking Description: The allocation to intervention or control groups is not random, but separated according to sports schools. This is the only way to ensure that there is no overlapping of training.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): All players in the intervention group will complete the targeted muscle and technique training integrated into their handball training. There will be a training of the coaches on site, who assess the training of the intervention group during the entire period and document the participation of the players accordingly.
  Interventions: Other: Muscle and technique training
- Control group (No Intervention): Players in the control group only continue their regular handball training.

INTERVENTIONS:
Other: Muscle and technique training — The strength training consists of three exercises (clam shell, side plank, calf raises) with an progressive overload after two to three weeks to ensure a continuous muscle stimulation. The technique training consists of different cutting variations with a focus on forefoot landings and conscious control of the knee to avoid high knee valgus movement and KAM respectively.
  Arms: Intervention group

SUMMARY:
Anterior cruciate ligament (ACL) injury constitutes the largest problem in female elite ball/team sport today, due to its relatively high incidence and serious short- and long-term consequences. Especially in handball, these injuries typically occur in actions that are essential for the game, i.e. landings and cutting maneuvers, imposing a challenge for risk reduction strategies. Although knowledge about risk factors is constantly increasing and ACL injury prevention programs have been successful in reducing injuries in rigorous scientific study settings, the real-world injury incidence remains high, and even continues to increase. The purpose of this explorative intervention study is to assess the effect of an eight-week strength and technique training in female handball players and its influence on ACL-specific risk factors, especially knee abduction moment (KAM). The results are compared with a control group that did not do the specially designed technique/muscle training.

DETAILED DESCRIPTION:
BACKGROUND:

ACL injuries are the number one problem in female elite ball/team sports due to its relatively high incidence and serious short- and long-term consequences. Typically injuries occur in actions that are essential for the game, i.e. landings and cutting maneuvers, imposing a challenge for risk reduction strategies.

The consequences of an ACL injury are manifold for the players. They not only reduce quality of life but also lead to a loss of social contacts due to missed training sessions what can be difficult, especially for younger players. Additionally, there are serious long-term consequences with a high likelihood of early osteoarthritis, lasting pain and disability. Also the risk of suffering a second ACL injury after returning to sport is high. In fact, as many as 20-30% of female players returning to play after an ACL injury end up with a new ACL injury in the same or contralateral knee, which makes prevention of a first injury even more important.

Video analyses of ACL injuries strongly suggest that biomechanics is important in injury causation. Novel model-based image-matching techniques have shown that valgus movement occurs shortly after initial contact of the foot with the ground. This implies that knee abduction loading is a likely causative factor. Still, video-based methods have limitations in their accuracy and detail level. To address this knowledge gap, the Oslo Sports Trauma Research Center has carried out the world's largest prospective risk factor study on ACL injuries to date-with multiple data collections between 2007 and 2014.

The most recent analyses indicate that there are clear associations between biomechanics of cutting maneuvers and injury risk. Specifically knee abduction moments seems to be greater in players who later go on to sustain an injury and can be affected by the players' cutting technique variables (width of cut, hip abduction, foot rotation, torso movement/rotation, hip rotation, knee valgus, knee flexion, cutting angle, cutting time, approach speed). These findings may simply reflect that injuries take place in cutting maneuvers and underline the importance of investigating such maneuvers, which closely mimic the real-life setting.

Resulting, there are several different cutting technique strategies, where some strategies may lead to a higher risk for ACL injury while others seem to reduce the risk of injury. Especially landing on the forefoot, rather than on the heel, showed to reduce knee abduction moments by 13% and it was found that a narrow cut, rather than a wide-stance cut, reduced knee abduction moments by 17%.

Based on this knowledge, the investigators want to find out whether it is possible to reduce the players' knee loading, especially reduce KAM, through influencing known risk factors for ACL injuries using a specially designed eight-week muscle and technique training.

AIMS:

The aim of this feasibility study is to assess the effect of an eight-week strength and technique training in female handball players on known risk factors for ACL injuries, especially the knee abduction moment (KAM).

STUDY DESIGN AND METHODS:

To recruit participants, the investigators will contact sports schools in and around Oslo that have a focus on handball. The study is a feasibility study with the aim of finding out whether a targeted, eight-week muscle and technique training based on known ACL-injury risk factors can have a positive influence on their reduction.

At baseline, there will be a 3D motion analysis of all participants (25 in the intervention group, 25 in the control group) performing sidestep cuttings (3 trials per side) in the biomechanical laboratory of the Norwegian School of Sport Sciences (NiH) in Oslo, as well as a strength measurement.

Although a variety of biomechanical data (centre of mass, specific joint positions, cutting width, speed, etc.) is collected as part of the analysis, the focus is on ACL-specific risk factors such as forefoot landing and KAM. The strength test focuses on hip abduction and external rotation, as well as a measurement of the posterior calf muscles.

All players in the intervention group will complete the targeted muscle and technique training integrated into their handball training, while players in the control group only continue their regular handball training. There will be a training of the coaches on site, who assess the training of the intervention group during the entire period and document the participation of the players accordingly.

The strength training consists of three exercises (clam shell, side plank, calf raises) with an progressive overload after two to three weeks to ensure a continuous muscle stimulation. The technique training consists of different cutting variations with a focus on forefoot landings and conscious control of the knee to avoid high knee valgus movement and KAM respectively.

The allocation to intervention or control groups is not random, but separated according to sports schools. This is the only way to ensure that there is no overlapping of training. After a eight-week intervention period, all participants will perform a post-test including the same previous mentioned outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Female handball players between the ages of 15 and 18 who go to a sports school in Oslo
* Consent by the players, in the case of age below 16 years by their parents
* Match fitness on test day

Exclusion Criteria:

- History of ACL injury in the last 6 months before baseline testing

Ages: 15 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — ACL injury risk is higher in female handball players. Therefore the investigators want to investigate especially this vulnerable group.
Enrollment: 50 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Knee Abduction Moment (KAM) | Baseline, second testing 8-10 weeks later
  Peak Knee Abduction Moment (KAM) within the first 100ms after initial contact (IC) of the foot. A known risk factor for ACL injury.

SECONDARY OUTCOMES:
Cutting technique factors. These may affect the main outcome variable, but also performance | Baseline, follow-up 8-10 weeks later
  Cutting angle (°), approach speed (m/s), knee valgus (°), foot strike angle (°), foot rotation (°), width of cut (cm), hip abduction angle (°), torso rotation (°)
Strength factors. These may affect the main outcome variable, but also performance | Baseline, follow-up 8-10 weeks later
  Isometric hip abduction force (N), isometric hip external rotation force (N), isometric plantar flexion force (N)
Performance in a timed run-and-cut task. Run 5 m forward, turn 180 degrees and run back 5 m. | Baseline, follow-up 8-10 weeks later
  Total time Time 2,5-5m Time 5m - back to start
Player/trainer knowledge and motivation, implementation likelihood | 2-3 months after the follow-up
  Measured through questionnaires and Interviews

CONTACTS AND LOCATIONS:
Locations (1):
- Norwegian School of Sport Sciences, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alentorn-Geli E, Mendiguchia J, Samuelsson K, Musahl V, Karlsson J, Cugat R, Myer GD. Prevention of anterior cruciate ligament injuries in sports. Part I: systematic review of risk factors in male athletes. Knee Surg Sports Traumatol Arthrosc. 2014 Jan;22(1):3-15. doi: 10.1007/s00167-013-2725-3. Epub 2013 Oct 25. PMID 24385003
- [Background] Ardern CL, Ekas G, Grindem H, Moksnes H, Anderson A, Chotel F, Cohen M, Forssblad M, Ganley TJ, Feller JA, Karlsson J, Kocher MS, LaPrade RF, McNamee M, Mandelbaum B, Micheli L, Mohtadi N, Reider B, Roe J, Seil R, Siebold R, Silvers-Granelli HJ, Soligard T, Witvrouw E, Engebretsen L. 2018 International Olympic Committee consensus statement on prevention, diagnosis and management of paediatric anterior cruciate ligament (ACL) injuries. Knee Surg Sports Traumatol Arthrosc. 2018 Apr;26(4):989-1010. doi: 10.1007/s00167-018-4865-y. Epub 2018 Feb 17. PMID 29455243
- [Background] Ardern CL, Taylor NF, Feller JA, Webster KE. Fifty-five per cent return to competitive sport following anterior cruciate ligament reconstruction surgery: an updated systematic review and meta-analysis including aspects of physical functioning and contextual factors. Br J Sports Med. 2014 Nov;48(21):1543-52. doi: 10.1136/bjsports-2013-093398. Epub 2014 Aug 25. PMID 25157180
- [Background] Benjaminse A, Welling W, Otten B, Gokeler A. Novel methods of instruction in ACL injury prevention programs, a systematic review. Phys Ther Sport. 2015 May;16(2):176-86. doi: 10.1016/j.ptsp.2014.06.003. Epub 2014 Jun 19. PMID 25042094
- [Background] Dempsey AR, Lloyd DG, Elliott BC, Steele JR, Munro BJ. Changing sidestep cutting technique reduces knee valgus loading. Am J Sports Med. 2009 Nov;37(11):2194-200. doi: 10.1177/0363546509334373. Epub 2009 Jun 9. PMID 19509415
- [Background] Dempsey AR, Lloyd DG, Elliott BC, Steele JR, Munro BJ, Russo KA. The effect of technique change on knee loads during sidestep cutting. Med Sci Sports Exerc. 2007 Oct;39(10):1765-73. doi: 10.1249/mss.0b013e31812f56d1. PMID 17909404
- [Background] Filbay SR, Ackerman IN, Russell TG, Macri EM, Crossley KM. Health-related quality of life after anterior cruciate ligament reconstruction: a systematic review. Am J Sports Med. 2014 May;42(5):1247-55. doi: 10.1177/0363546513512774. Epub 2013 Dec 6. PMID 24318609
- [Background] Fox AS. Change-of-Direction Biomechanics: Is What's Best for Anterior Cruciate Ligament Injury Prevention Also Best for Performance? Sports Med. 2018 Aug;48(8):1799-1807. doi: 10.1007/s40279-018-0931-3. PMID 29721837
- [Background] Grindem H, Snyder-Mackler L, Moksnes H, Engebretsen L, Risberg MA. Simple decision rules can reduce reinjury risk by 84% after ACL reconstruction: the Delaware-Oslo ACL cohort study. Br J Sports Med. 2016 Jul;50(13):804-8. doi: 10.1136/bjsports-2016-096031. Epub 2016 May 9. PMID 27162233
- [Background] Havens KL, Sigward SM. Cutting mechanics: relation to performance and anterior cruciate ligament injury risk. Med Sci Sports Exerc. 2015 Apr;47(4):818-24. doi: 10.1249/MSS.0000000000000470. PMID 25102291
- [Background] Huang YL, Jung J, Mulligan CMS, Oh J, Norcross MF. A Majority of Anterior Cruciate Ligament Injuries Can Be Prevented by Injury Prevention Programs: A Systematic Review of Randomized Controlled Trials and Cluster-Randomized Controlled Trials With Meta-analysis. Am J Sports Med. 2020 May;48(6):1505-1515. doi: 10.1177/0363546519870175. Epub 2019 Aug 30. PMID 31469584
- [Background] Koga H, Nakamae A, Shima Y, Iwasa J, Myklebust G, Engebretsen L, Bahr R, Krosshaug T. Mechanisms for noncontact anterior cruciate ligament injuries: knee joint kinematics in 10 injury situations from female team handball and basketball. Am J Sports Med. 2010 Nov;38(11):2218-25. doi: 10.1177/0363546510373570. Epub 2010 Jul 1. PMID 20595545
- [Background] Kristianslund E, Bahr R, Krosshaug T. Kinematics and kinetics of an accidental lateral ankle sprain. J Biomech. 2011 Sep 23;44(14):2576-8. doi: 10.1016/j.jbiomech.2011.07.014. Epub 2011 Aug 6. PMID 21824618
- [Background] Kristianslund E, Faul O, Bahr R, Myklebust G, Krosshaug T. Sidestep cutting technique and knee abduction loading: implications for ACL prevention exercises. Br J Sports Med. 2014 May;48(9):779-83. doi: 10.1136/bjsports-2012-091370. Epub 2012 Dec 20. PMID 23258848
- [Background] Kristianslund E, Krosshaug T, Mok KM, McLean S, van den Bogert AJ. Expressing the joint moments of drop jumps and sidestep cutting in different reference frames--does it matter? J Biomech. 2014 Jan 3;47(1):193-9. doi: 10.1016/j.jbiomech.2013.09.016. Epub 2013 Oct 11. PMID 24161796
- [Background] Krosshaug T, Steffen K, Kristianslund E, Nilstad A, Mok KM, Myklebust G, Andersen TE, Holme I, Engebretsen L, Bahr R. Screening Tests for ACL Injury: Response. Am J Sports Med. 2016 Jun;44(6):NP26-7. doi: 10.1177/0363546516651046. No abstract available. PMID 27252550
- [Background] Krosshaug T, Steffen K, Kristianslund E, Nilstad A, Mok KM, Myklebust G, Andersen TE, Holme I, Engebretsen L, Bahr R. The Vertical Drop Jump Is a Poor Screening Test for ACL Injuries in Female Elite Soccer and Handball Players: A Prospective Cohort Study of 710 Athletes. Am J Sports Med. 2016 Apr;44(4):874-83. doi: 10.1177/0363546515625048. Epub 2016 Feb 11. PMID 26867936
- [Background] Lie MM, Risberg MA, Storheim K, Engebretsen L, Oiestad BE. What's the rate of knee osteoarthritis 10 years after anterior cruciate ligament injury? An updated systematic review. Br J Sports Med. 2019 Sep;53(18):1162-1167. doi: 10.1136/bjsports-2018-099751. Epub 2019 Apr 1. PMID 30936063
- [Background] Mok KM, Bahr R, Krosshaug T. Reliability of lower limb biomechanics in two sport-specific sidestep cutting tasks. Sports Biomech. 2018 Jun;17(2):157-167. doi: 10.1080/14763141.2016.1260766. Epub 2017 Mar 10. PMID 28281390
- [Background] Myklebust G, Bahr R, Nilstad A, Steffen K. Knee function among elite handball and football players 1-6 years after anterior cruciate ligament injury. Scand J Med Sci Sports. 2017 May;27(5):545-553. doi: 10.1111/sms.12842. Epub 2017 Mar 8. PMID 28107551
- [Background] Pairot-de-Fontenay B, Willy RW, Elias ARC, Mizner RL, Dube MO, Roy JS. Running Biomechanics in Individuals with Anterior Cruciate Ligament Reconstruction: A Systematic Review. Sports Med. 2019 Sep;49(9):1411-1424. doi: 10.1007/s40279-019-01120-x. PMID 31102111
- [Background] Pasanen K, Rossi MT, Parkkari J, Heinonen A, Steffen K, Myklebust G, Krosshaug T, Vasankari T, Kannus P, Avela J, Kulmala JP, Perttunen J, Kujala UM, Bahr R. Predictors of lower extremity injuries in team sports (PROFITS-study): a study protocol. BMJ Open Sport Exerc Med. 2015 Dec 11;1(1):e000076. doi: 10.1136/bmjsem-2015-000076. eCollection 2015. PMID 27900143
- [Background] Petushek EJ, Sugimoto D, Stoolmiller M, Smith G, Myer GD. Evidence-Based Best-Practice Guidelines for Preventing Anterior Cruciate Ligament Injuries in Young Female Athletes: A Systematic Review and Meta-analysis. Am J Sports Med. 2019 Jun;47(7):1744-1753. doi: 10.1177/0363546518782460. Epub 2018 Jul 12. PMID 30001501
- [Background] Sharir R, Rafeeuddin R, Staes F, Dingenen B, George K, Vanrenterghem J, Robinson MA. Mapping current research trends on anterior cruciate ligament injury risk against the existing evidence: In vivo biomechanical risk factors. Clin Biomech (Bristol). 2016 Aug;37:34-43. doi: 10.1016/j.clinbiomech.2016.05.017. Epub 2016 Jun 2. PMID 27286556
- [Background] Steffen K, Nilstad A, Kristianslund EK, Myklebust G, Bahr R, Krosshaug T. Association between Lower Extremity Muscle Strength and Noncontact ACL Injuries. Med Sci Sports Exerc. 2016 Nov;48(11):2082-2089. doi: 10.1249/MSS.0000000000001014. PMID 27327027
- [Background] Sugimoto D, Myer GD, Foss KD, Hewett TE. Specific exercise effects of preventive neuromuscular training intervention on anterior cruciate ligament injury risk reduction in young females: meta-analysis and subgroup analysis. Br J Sports Med. 2015 Mar;49(5):282-9. doi: 10.1136/bjsports-2014-093461. Epub 2014 Dec 1. PMID 25452612
- [Background] Whittaker JL, Woodhouse LJ, Nettel-Aguirre A, Emery CA. Outcomes associated with early post-traumatic osteoarthritis and other negative health consequences 3-10 years following knee joint injury in youth sport. Osteoarthritis Cartilage. 2015 Jul;23(7):1122-9. doi: 10.1016/j.joca.2015.02.021. Epub 2015 Feb 26. PMID 25725392